CLINICAL TRIAL: NCT02372799
Title: A Multicenter, Double-blind, Placebo- and Active-Controlled Parallel-Group Evaluation of the Safety and Efficacy of Vilazodone in Pediatric Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Vilazodone in Pediatric Patients With Major Depressive Disorder (VLZ-MD-22)
Acronym: VLZ-MD-22
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VLZ-MD-22
Record Dates: First submitted 2015-02-21; First posted 2015-02-26 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vilazodone Hydrochloride; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vilazodone (Experimental): Vilazodone tablets, 5mg, 10mg and 20mg. Oral administration, once per day.
  Interventions: Drug: Vilazodone
- Placebo (Placebo Comparator): Dose-matched placebo tablets or capsules, oral administration, once per day.
  Interventions: Drug: Placebo
- Fluoxetine (Active Comparator): Fluoxetine capsules, 10mg and 20 mg. Oral administration, once per day.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Vilazodone
  Other Names: Viibryd
  Arms: Vilazodone
Drug: Placebo
  Arms: Placebo
Drug: Fluoxetine
  Other Names: Prozac
  Arms: Fluoxetine

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of vilazodone compared with placebo in pediatric outpatients (7-17 years of age) with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female outpatients between 7-17 years of age
* Primary diagnosis of Major Depressive Disorder (MDD)
* Children's Depression Rating Scale-Revised (CDRS-R) score of 40 or greater
* Clinical Global Impressions-Severity (CGI-S) score of 4 or greater

Exclusion Criteria:

* Current (past 3 months) principal Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR) based diagnosis of an axis disorder other than major depressive disorder (MDD) that is the primary focus of treatment.
* History of suicidal behavior, or requires precaution against suicide
* Not generally healthy medical condition
* Seizure disorder

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 473 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily McCusker, PhD, Study Director — Forest Research Institute, an affiliate of Allergan plc.
Locations (60):
- United States (58):
  - Alliance Clinical Research, Birmingham, Alabama
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Woodland International Research Group, INC, Little Rock, Arkansas
  - CITrials - Bellflower, Bellflower, California
  - ATP Clinical Research, Costa Mesa, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - PCSD - Feighner Research, San Diego, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Hartford Hospital, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Palm Springs Research, LLC, Hialeah, Florida
  - IMIC Inc., Homestead, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Osceola Mental Health dba Park Place Behavioral Health Care, Kissimmee, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlantic Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - Neuroscience Research Institute Inc., Oak Park, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Hugo W Moser Research Institute at Kennedy Krieger, Inc., Baltimore, Maryland
  - Pharmsite Research Inc., Baltimore, Maryland
  - NeuroScientific Insights, Rockville, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - BioScience Research LLC, Mount Kisco, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Finger Lakes Clinical research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Haidar Almhana Nieding LLC, Avon Lake, Ohio
  - Neuro-Behavioral Clinical Research, Inc, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Psychiatry, Cleveland, Ohio
  - Ohio State Univ. Dept of Psychiatry, Columbus, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Research Strategies of Memphis LLC, Memphis, Tennessee
  - FutureSearch Clinical trials, Inc., Austin, Texas
  - BioBehavioral Research of Austin, PC, Austin, Texas
  - University of TX Southwestern Medical Ctr, Dallas, Texas
  - Bayou City Research Ltd, Houston, Texas
  - Houston Endoscopy and Research Ctr, Houston, Texas
  - Research Across America, Plano, Texas
  - Focus and Balance, San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Ericksen Research and Development, Clinton, Utah
  - UVA Center for Psychopharmacology Research in Youth, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Everett, Washington
- Canada (2):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Paediatric Sleep Research Inc, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization and treatment assignment were based on a randomization scheme prepared by Allergan Biostatistics prior to the start of the study
Groups:
- Vilazodone: Vilazodone tablets 15-30 mg. Oral administration, once per day.
- Fluoxetine: Fluoxetine capsules 20 mg. Oral administration, once per day.
Period: Treatment Period
Arm/Group | Placebo | Vilazodone | Fluoxetine
Started | 186 | 187 | 97
Completed | 152 | 155 | 82
Not Completed | 34 | 32 | 15
Not completed — Adverse Event | 3 | 10 | 6
Not completed — Insufficient therapeutic response | 2 | 2 | 0
Not completed — Withdrawal by Subject | 10 | 10 | 2
Not completed — Lost to Follow-up | 11 | 5 | 3
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Non-compliance with study drug | 4 | 4 | 4
Not completed — Miscellaneous Reasons | 1 | 1 | 0
Period: Down-taper Period
Arm/Group | Placebo | Vilazodone | Fluoxetine
Started | 152 | 159 | 82
Completed | 151 | 157 | 80
Not Completed | 1 | 2 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Population will consist of all patients in the Randomized Population who received at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilazodone | Fluoxetine | Total
Number analyzed (Participants) | 186 | 187 | 97 | 470
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13 (2.9) | 13 (2.9) | 13.2 (2.8) | 13 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  7-11 | 61 | 55 | 30 | 146
  12-17 | 125 | 132 | 67 | 324
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 126 | 51 | 283
  Male | 80 | 61 | 46 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 25 | 12 | 64
  Not Hispanic or Latino | 159 | 162 | 85 | 406
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 118 | 121 | 60 | 299
  Black or African American | 57 | 58 | 30 | 145
  Asian | 5 | 1 | 1 | 7
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  Other | 5 | 5 | 5 | 15
  Missing | 0 | 0 | 1 | 1
Weight [Mean (Standard Deviation); unit: kg] | 59.13 (24.29) | 61.35 (24.79) | 59.38 (21.14) | 60.07 (23.86)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 23.31 (6.85) | 24.25 (7.58) | 23.48 (6.66) | 23.72 (7.11)
CDRS-R total score [Mean (Standard Deviation); unit: units on a scale] — The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 133 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood. Population: The CDRS-R total score is provided at baseline for the Intent to Treat study population, which comprises the 465 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
  units on a scale
    number analyzed (Participants) | 182 | 186 | 97 | 465
    (all) | 57.3 (9.2) | 58.3 (9.2) | 58 (8.8) | 57.8 (9.1)
CGI-S score [Mean (Standard Deviation); unit: Units on a Scale] — The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated instrument used to rate the severity of the patient's current state of mental illness compared with the clinician's total experience with patients with major depressive disorder (MDD). The severity of the patient's MDD was rated on a scale from 1 to 7, with 1 indicating a normal state and 7 indicating a patient who is among the most extremely ill patients. Population: The CGI-S score is provided at baseline for the Intent to Treat study population, which comprises the 465 patients in the Safety Population who had a baseline and at least 1 postbaseline assessment of the CDRS-R total score.
  Units on a Scale
    number analyzed (Participants) | 182 | 186 | 97 | 465
    (all) | 4.6 (0.6) | 4.7 (0.6) | 4.6 (0.6) | 4.6 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Children's Depression Rating Scale-Revised (CDRS-R) Total Score
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 133 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood.
Time Frame: From Baseline to Week 8
Population: The Intent-to-Treat (ITT) Population will consist of all patients in the Safety Population who had baseline and at least 1 postbaseline assessment of the Children's Depression Rating Scale-Revised (CDRS-R) total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vilazodone | Fluoxetine
Number analyzed (Participants) | 182 | 186 | 97
units on a scale | -20.32 (0.983) | -20.72 (0.977) | -22.71 (1.320)
Statistical Analysis 1: Comparison: Placebo vs Vilazodone; Test type: Superiority; p = 0.7662, MMRM; LSMD = -0.40, 95% CI 2-sided [-3.08 to 2.27]
Statistical Analysis 2: Comparison: Placebo vs Fluoxetine; Test type: Superiority; p = 0.1433, MMRM; LSMD = -2.39, 95% CI 2-sided [-5.60 to 0.81]

2. Secondary Outcome: Change in Clinical Global Impressions-Severity (CGI-S) Score
Description: The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated instrument used to rate the severity of the patient's current state of mental illness compared with the clinician's total experience with patients with major depressive disorder (MDD). The severity of the patient's MDD was rated on a scale from 1 to 7, with 1 indicating a normal state and 7 indicating a patient who is among the most extremely ill patients.
Time Frame: From Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vilazodone | Fluoxetine
Number analyzed (Participants) | 182 | 186 | 97
units on a scale | -1.52 (0.097) | -1.57 (0.096) | -1.72 (0.130)
Statistical Analysis 1: Comparison: Placebo vs Vilazodone; Test type: Superiority; p = 0.7387, MMRM; LSMD = -0.04, 95% CI 2-sided [-0.31 to 0.22]
Statistical Analysis 2: Comparison: Placebo vs Fluoxetine; Test type: Superiority; p = 0.2158, MMRM; LSMD = -0.20, 95% CI 2-sided [-0.52 to 0.12]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the participant's signing of the Informed Consent Forum until 30 days after the last does of study treatment, spanning a period of 10 to 13 weeks.
Arm/Group | Placebo | Vilazodone | Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/186 | 0/187 | 0/97
Serious Adverse Events (participants affected / at risk) | 1/186 | 0/187 | 6/97
Other Adverse Events (participants affected / at risk) | 54/186 | 97/187 | 27/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Vilazodone (N=187) | Fluoxetine (N=97)
Croup infectious (Infections and infestations) | 1 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=186) | Vilazodone (N=187) | Fluoxetine (N=97)
Nausea (Gastrointestinal disorders) | 13 | 40 | 6
Vomiting (Gastrointestinal disorders) | 7 | 24 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 16 | 2
Abdominal pain upper (Gastrointestinal disorders) | 6 | 13 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 5
Headache (Nervous system disorders) | 31 | 24 | 10
Somnolence (Nervous system disorders) | 4 | 12 | 2
Dizziness (Nervous system disorders) | 5 | 10 | 2
Insomnia (Psychiatric disorders) | 3 | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study are the property of the sponsor. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and the sponsor and will follow sponsor's standard operating procedures on publications.

DOCUMENTS (2):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/99/NCT02372799/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT02372799/SAP_001.pdf